CLINICAL TRIAL: NCT05976412
Title: Prospective Randomized Controlled Study on Precision Irradiation of Regional Lymph Node for Clinical High-risk pN0 Breast Cancer
Brief Title: Regional Lymph Node Irradiation for High-risk pN0 Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, JIAYI CHEN, Prof, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023（148）
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RNI group (Experimental)
  Interventions: Radiation: Regional lymph node radiotherapy; Radiation: chest/whole breast irradiation
- non-RNI group (Placebo Comparator)
  Interventions: Radiation: chest/whole breast irradiation

INTERVENTIONS:
Radiation: Regional lymph node radiotherapy — Regional lymph node radiotherapy
  Arms: RNI group
Radiation: chest/whole breast irradiation — chest/whole breast irradiation

SUMMARY:
This study is a non blind, randomized controlled study, whose hypothesis was that chest wall/whole breast combined regional lymph node radiotherapy can improve the 5-year disease-free survival rate of clinical high-risk pN0 breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Voluntarily participate and sign an informed consent form; Age>18 years old, female； received radical surgery for breast cancer, including breast conservation surgery or mastectomy, combined with Sentinel lymph node biopsy or axillary lymph node dissection； Invasive cancer, postoperative axillary lymph node negative, with pathological staging of T1-3N0M0 stage (Stage IA, IIA, IIB)； including two or more high-risk factors based on four clinical high-risk recurrence factors [tumor size (>2cm), tumor site (medial and central quadrants), Ki-67 level (>14%), and vascular status (positive)]; KPS ≥ 80, estimated survival time >5 years; Complete healing of Surgical incision, no incision infection, etc; Reproductive period women should undergo contraception for at least one month before study, and promise to use contraception throughout the entire study period and continue until the specified time after the end of the study

Exclusion Criteria:

Pregnant or lactating women; Received neoadjuvant therapy; with serious non neoplastic medical complications that affect the implementation of radiotherapy; History of malignant tumor in the past 5 years (excluding previous lobular Carcinoma in situ, skin Basal-cell carcinoma, skin Carcinoma in situ, cervical Carcinoma in situ and lung Carcinoma in situ); Simultaneous contralateral breast cancer; Previous history of neck, chest, or ipsilateral axillary radiotherapy; Active collagen vascular disease; distant metastasis confirmed by pathology or imaging;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1355 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2031-05-31 (Estimated); Study Completion 2031-05-31 (Estimated)

PRIMARY OUTCOMES:
5 year disease free survival rate | 5 year
  Disease free survival rate from randomization to 5 years after radiotherapy

SECONDARY OUTCOMES:
5 year local reginal recurrence rate | 5 year
  The proportion of local or regional recurrence from randomization to 5 years after radiotherapy
5 year distant metastases rate | 5 year
  The proportion of distant metastases occurring 5 years after radiotherapy
5 year overall survival rate | 5 year
  The proportion of death occurring 5 years after radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai jiaotong univestigy school of medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided